CLINICAL TRIAL: NCT05880992
Title: Trimodal Prehabilitation in Colorectal Cancer Patients: a Feasibility Pilot
Brief Title: Trimodal Prehabilitation in Colorectal Cancer Patients
Acronym: PrehabCRC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan Leitch (Other)
Responsible Party: Sponsor-Investigator, Jordan Leitch, Staff Physician, Assistant Professor, Department of Anesthesiology and Perioperative Medicine, Queen's University
Organization: Queen's University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PrehabCRC
Record Dates: First submitted 2023-05-16; First posted 2023-05-30 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Exercise; Nutritional Status; Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progress Check (Other): This arm will include pre- and post-prehabilitation questionnaires as well as twice weekly progress checks by the research assistant to check on participant progress, answer questions and provide accountability and motivation.
  Interventions: Behavioral: Exercise; Dietary Supplement: Nutrition; Behavioral: Mindfulness
- No Progress Check (Other): This arm will include only pre- and post-prehabilitation questionnaires.
  Interventions: Behavioral: Exercise; Dietary Supplement: Nutrition; Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Exercise — Aerobic and Strength exercises (equipment free, simple, modifiable)
Dietary Supplement: Nutrition — Counselling on daily protein target of 1.2 g/kg as well as supplementation with protein shake (provided)
Behavioral: Mindfulness — Deep (box) breathing completing in the morning, evening and as needed.

SUMMARY:
The goal of this clinical pilot is to determine the feasibility of implementing trimodal prehabilitation within the current perioperative infrastructure in patients having major colorectal surgery for resection of a cancer (CRC). Trimodal prehabilitation includes exercise, nutrition and mindfulness coaching and support which has been shown to improve physical status, mental preparation and to reduce loss of lean body mass in CRC patients. The primary questions this study aims to answer are: Is delivery of trimodal prehabilitation feasible within our current perioperative infrastructure and does prehabilitation impact outcomes in these patients? Researchers will compare this newly recruited prehabilitation cohort to a historical cohort of patients who did not receive prehabilitation in terms of mortality, length of stay, complications, readmissions, emergency department visits and non-home discharge.

DETAILED DESCRIPTION:
Fifty patients aged 18 years or greater booked to undergo major colorectal surgery (colectomy, low anterior resection or abdominoperineal resection) will be enrolled from June to August 2023 from the colorectal cancer (CRC) clinic at Kingston Health Sciences Centre in Kingston, Ontario. The CRC nurse navigator will identify new CRC diagnoses coming into clinic and will alert the research team. A research assistant will attend the CRC clinic when potentially eligible patients are booked and will approach regarding recruitment into the study. Exclusion criteria will include refusal to participate in study and inability to understand questionnaires and participate in psychological assessments in English. Once recruited to study, the research assistant will give the patient the prehabilitation resources (including a prescription for aerobic and strength exercises to be completed each week, 36 Premier Protein shakes (30g protein, 150 calories per shake) and a handout describing deep breathing exercises) and arrange a time with the patient to complete baseline questionnaires and deliver prehabilitation consultation. The rationale for delaying this initial consultation is to prevent overwhelming patients with information after receiving a new cancer diagnosis. Patients will have a prehabilitation study consultation including completion of three questionnaires: self-assessment of physical activity (CHAMPS), nutritional screening (CNST) and health care related quality of life (SF-36). Patients will then be given all prehabilitation education and counselling.

Study patients will participate in a trimodal prehabilitation program (including exercise, nutrition and mindfulness goals) prior to surgery, and will be randomized into two groups: 1) Prehabilitation with twice-weekly progress checks (adherence to prehabilitation program) and 2) Prehabilitation without progress checks. Both groups of patients will complete daily activity trackers to document exercise completion, protein drink consumption and deep breathing exercises. One week prior to surgery, a research assistant will contact all participants and conduct CHAMPS, CNST and SF-36 as well as collect feasibility outcomes including weeks available for prehabilitation before surgery, satisfaction with prehabilitation program and adherence to program (participating in phone calls, completing exercises, daily protein shake (30g) and mindfulness exercise). Groups that are designated as including progress checks will be called by a research assistant twice per week to check in on progress regarding all components of prehabilitation program (adherence, compliance, issues).

An additional analysis will be performed comparing the 50 patients from this feasibility pilot (prehabilitation group) to the previous 50 patients booked for major colorectal surgery (standard care group) using existing data from the colorectal database. These groups will be assessed for secondary outcomes including mortality, length of stay, emergency department visits, readmissions, major complications and non-home discharge. This pilot study will guide the development of a larger study to assess the delivery of prehabilitation and rehabilitation after major colorectal surgery utilizing CloudDX, software that can be programmed to deliver reminders, surveys and important information to assist with adherence to the prehabilitation regimen. In addition, these future studies will utilize remote vital sign monitoring via CloudDX to collect important biometric data to richen the interpretation of the effects of prehabilitation on this patient population.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* major colorectal surgery (colectomy, low anterior resection or abdominoperineal resection)

Exclusion Criteria:

* refusal to participate in study
* inability to understand questionnaires and participate in psychological assessments in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Retention rate | Four to six weeks prior to surgery
  Rate of participants who completed entire duration of prehabilitation, regardless of components performed
Recruitment rate | Four to six weeks prior to surgery
  Number of patients booked for surgery compared to the number of overall patients booked for surgery during the study timeframe.
Exercise completion rate | Four to six weeks prior to surgery
  Percentage of strength exercises completed and percentage of aerobic exercise completed
Nutrition compliance rate | Four to six weeks prior to surgery
  Percentage of days protein shake was consumed
Mindfulness compliance rate | Four to six weeks prior to surgery
  Percentage of deep breathing exercises performed
Adherence rate | Four to six weeks prior to surgery
  Percentage of all components of prehabilitation completed by participants

SECONDARY OUTCOMES:
All-cause Mortality | 30 days after surgery
  Number of participants who died from any cause
Readmission to hospital | 30 days after surgery
  Number of participants who were re-admitted to hospital
Presentation to emergency department | 30 days after surgery
  Number of participants who presented to the emergency department
Non-home discharge | 30 days after surgery
  Number of participants discharged to a non-home location
Major complications | 30 days after surgery
  Rate of surgical site infection and major bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Leitch, Principal Investigator — Queen's University
Locations (1):
- Kingston Health Sciences Centre, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bojesen RD, Jorgensen LB, Grube C, Skou ST, Johansen C, Dalton SO, Gogenur I. Fit for Surgery-feasibility of short-course multimodal individualized prehabilitation in high-risk frail colon cancer patients prior to surgery. Pilot Feasibility Stud. 2022 Jan 21;8(1):11. doi: 10.1186/s40814-022-00967-8. PMID 35063042
- [Background] Chmelo J, Phillips AW, Greystoke A, Charman SJ, Avery L, Hallsworth K, Welford J, Cooper M, Sinclair RCF. A feasibility trial of prehabilitation before oesophagogastric cancer surgery using a multi-component home-based exercise programme: the ChemoFit study. Pilot Feasibility Stud. 2022 Aug 9;8(1):173. doi: 10.1186/s40814-022-01137-6. PMID 35945625
- [Background] Gillis C, Fenton TR, Sajobi TT, Minnella EM, Awasthi R, Loiselle SE, Liberman AS, Stein B, Charlebois P, Carli F. Trimodal prehabilitation for colorectal surgery attenuates post-surgical losses in lean body mass: A pooled analysis of randomized controlled trials. Clin Nutr. 2019 Jun;38(3):1053-1060. doi: 10.1016/j.clnu.2018.06.982. Epub 2018 Jul 9. PMID 30025745
- [Background] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535
- [Background] Martin D, Besson C, Pache B, Michel A, Geinoz S, Gremeaux-Bader V, Larcinese A, Benaim C, Kayser B, Demartines N, Hubner M. Feasibility of a prehabilitation program before major abdominal surgery: a pilot prospective study. J Int Med Res. 2021 Nov;49(11):3000605211060196. doi: 10.1177/03000605211060196. PMID 34851778
- [Background] McAdams-DeMarco MA, Ying H, Van Pilsum Rasmussen S, Schrack J, Haugen CE, Chu NM, Gonzalez Fernandez M, Desai N, Walston JD, Segev DL. Prehabilitation prior to kidney transplantation: Results from a pilot study. Clin Transplant. 2019 Jan;33(1):e13450. doi: 10.1111/ctr.13450. Epub 2018 Dec 21. PMID 30462375
- [Background] McIsaac DI, Gill M, Boland L, Hutton B, Branje K, Shaw J, Grudzinski AL, Barone N, Gillis C; Prehabilitation Knowledge Network. Prehabilitation in adult patients undergoing surgery: an umbrella review of systematic reviews. Br J Anaesth. 2022 Feb;128(2):244-257. doi: 10.1016/j.bja.2021.11.014. Epub 2021 Dec 16. PMID 34922735
- [Background] McIsaac DI, Hladkowicz E, Bryson GL, Forster AJ, Gagne S, Huang A, Lalu M, Lavallee LT, Moloo H, Nantel J, Power B, Scheede-Bergdahl C, van Walraven C, McCartney CJL, Taljaard M. Home-based prehabilitation with exercise to improve postoperative recovery for older adults with frailty having cancer surgery: the PREHAB randomised clinical trial. Br J Anaesth. 2022 Jul;129(1):41-48. doi: 10.1016/j.bja.2022.04.006. Epub 2022 May 17. PMID 35589429